CLINICAL TRIAL: NCT01553578
Title: The Efficacy of Healing Touch Versus Guided Imagery on Pain, Fatigue, Nausea, and Anxiety in Patients' Receiving Outpatient Chemotherapy
Brief Title: Healing Touch or Guided Imagery In Treating Pain, Fatigue, Nausea, and Anxiety in Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00018805; NCI-2012-00164 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 97511 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2012-03-09; First posted 2012-03-14 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Anxiety Disorder; Fatigue; Malignant Neoplasm; Nausea and Vomiting; Pain
MeSH Terms: conditions — Anxiety Disorders; Fatigue; Neoplasms; Nausea; Vomiting; Pain | interventions — Therapeutic Touch; Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (healing touch therapy) (Experimental): Patients receive 30 minutes of healing touch therapy consisting of magnetic clearing, pain drains, hands in motion/hands still and mind clearing.
  Interventions: Other: questionnaire administration; Procedure: therapeutic touch; Behavioral: management of therapy complications
- Arm B (guided imagery) (Experimental): Patients listen to guided imagery audiotapes for 30 minutes.
  Interventions: Other: questionnaire administration; Behavioral: management of therapy complications
- Arm C (standard care) (Active Comparator): Patients receive standard of care.
  Interventions: Other: questionnaire administration; Procedure: standard follow-up care

INTERVENTIONS:
Other: questionnaire administration — Ancillary studies
Procedure: therapeutic touch — Receive healing touch therapy
  Other Names: healing touch
  Arms: Arm A (healing touch therapy)
Behavioral: management of therapy complications — Receive healing touch therapy
  Other Names: complications of therapy, management of
  Arms: Arm A (healing touch therapy)
Behavioral: management of therapy complications — Receive guided imagery audiotapes
  Other Names: complications of therapy, management of
  Arms: Arm B (guided imagery)
Procedure: standard follow-up care — Receive standard care
  Arms: Arm C (standard care)

SUMMARY:
This randomized clinical trial studies healing touch or guided imagery in treating pain, fatigue, nausea, and anxiety in patients undergoing chemotherapy. Healing touch and guided imagery may help treat complications caused by chemotherapy. It is not yet known whether healing touch or guided imagery is more effective in treating pain, fatigue, nausea, and anxiety in patients undergoing chemotherapy

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the provision of healing touch or guided imagery during outpatient chemotherapy is associated with decreased pain, fatigue, nausea and anxiety when compared to standard outpatient treatment protocols.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM A: Patients receive 30 minutes of healing touch therapy comprising magnetic clearing, pain drains, hands in motion/hands still and mind clearing.

ARM B: Patients listen to guided imagery audiotapes for 30 minutes

ARM C: Patients receive standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at the outpatient chemotherapy area will be enrolled without consideration for type of cancer or chemotherapeutic agents to be used

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change scores for each patient on pain scale | Approximately 6 months
  Collected using a 10 point visual analog scale for pain, fatigue, nausea, and anxiety. Analyzed initially using descriptive statistics. Compared among the 3 groups using one-way analysis of variance (ANOVA) models and 2-sample t-tests.
Change scores for each patient on fatigue scale | Approximately 6 months
  Collected using a 10 point visual analog scale for pain, fatigue, nausea, and anxiety. Analyzed initially using descriptive statistics. Compared among the 3 groups using one-way analysis of variance (ANOVA) models and 2-sample t-tests.
Change scores for each patient on nausea scale | Approximately 6 months
  Collected using a 10 point visual analog scale for pain, fatigue, nausea, and anxiety. Analyzed initially using descriptive statistics. Compared among the 3 groups using one-way analysis of variance (ANOVA) models and 2-sample t-tests.
Change scores for each patient on anxiety scale | Approximately 6 months
  Collected using a 10 point visual analog scale for pain, fatigue, nausea, and anxiety. Analyzed initially using descriptive statistics. Compared among the 3 groups using one-way analysis of variance (ANOVA) models and 2-sample t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Hodges, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States